CLINICAL TRIAL: NCT05788887
Title: Postprandial Inflammatory and Metabolic Responses Induced by the Authentic Ladotyri Mytilinis PDO Cheese and Italian Parmesan PDO Cheese
Brief Title: Investigation of the Postprandial Response of Two Different PDO Cheeses on Metabolic Biomarkers
Acronym: LadotyriCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Aegean (Other)
Collaborators: E.Thimelis Dairy S.A. (Unknown)
Responsible Party: Principal Investigator, ANTONIOS KOUTELIDAKIS, Professor Antonios E. Koutelidakis, University of the Aegean
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BAP20060569
Record Dates: First submitted 2023-02-24; First posted 2023-03-29 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Ladotyri Mytilinis PDO cheese; Postprandial response

STUDY DESIGN:
Intervention Model Description: In the first trial period, participants in arm a consumed a meal containing 100g of white wheat bread and 80g of Italian Parmesan PDO cheese and arm b participants consumed a meal containing 100g of white wheat bread and 80g of Authentic Ladotyri Mytilinis PDO cheese. After a washout week participants consumed the meals, in reverse.
Who Masked: Participant
Masking Description: Only investigator knew the type of meal, consumed by each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The meal contained 100g of white wheat bread and 80g of Italian Parmesan PDO cheese.
  Interventions: Other: Control
- Intervention (Other): The meal contained 100g of white wheat bread and 80g of Authentic Ladotyri Mytilinis PDO cheese.
  Interventions: Other: Authentic Ladotyri Mytilinis PDO cheese

INTERVENTIONS:
Other: Authentic Ladotyri Mytilinis PDO cheese — Branding PDO cheese from Mytilini, purchasing by E.Thimelis Dairy S.A.
  Arms: Intervention
Other: Control — Branding Parmesan PDO cheese from Italy, supplied by LIDL Hellas
  Other Names: Italian Parmesan
  Arms: Control

SUMMARY:
The purpose of this study was the investigation of the postprandial metabolic responses, after the intake of a traditional, Ladotyri Mytilinis cheese, compared to corresponding responses after an Italian Parmesan cheese consumption, in healthy participants.

DETAILED DESCRIPTION:
A pilot cross-over, randomized and single-blinded, intervention-clinical trial was conducted, in ten healthy men and women subjects, aged eighteen to thirty years, after random allocation into the control and the intervention group, received a high-fat and carbohydrates meal, containing Ladotyri Mytilinis (the authentic nonrefrigerated recipe) or Italian Parmesan, PDO cheeses. After a washout week, participants consumed the same meals, conversely. Differences on postprandial responses of serum total, High Density Lipoprotein (HDL-), Low Density Lipoprotein (LDL-) cholesterol, glucose, triglycerides and uric acid levels, as well as of plasma total antioxidant capacity according to Ferric Reducing Antioxidant Power method, were determined between groups in fasting, thirty minutes, one and a half hour, and three hours after meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Willingness to join and complete the nutritional intervention

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Three-month nutritional supplement
* Age over 65 years or below 18 years
* Chronic diseases history
* Hemoglobin A1c - HbA1c > 5.7 %
* Abnormal Body Mass Index (BMI) (> 25 kg / m2)
* Abnormal hematological or biochemical profile (total cholesterol > 240 mg/dL, triglycerides > 250 mg/dL, glucose > 100 mg/dL)
* Alcohol overdose (> 40 g alcohol / day)
* Heavy smoking (> 10 cigarettes / day)
* Concurrent participation in another intervention study or unconsciousness in previous blood draws

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of Total Antioxidant Capacity at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Plasma antioxidant activity

SECONDARY OUTCOMES:
Changes from baseline of total Cholesterol at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum total cholesterol levels
Changes from baseline of High Density Lipoprotein cholesterol (HDL-) at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum High Density Lipoprotein levels
Changes from baseline of Low Density Lipoprotein cholesterol (LDL-) at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum High Density Lipoprotein levels
Changes from baseline of triglycerides at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum triglycerides levels
Changes from baseline of glucose at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum glucose levels
Changes from baseline of Uric Acid at 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum uric acid levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Aegean, Myrina, Greece

IPD SHARING:
Plan to Share IPD: No
No individual participant data are to be shared.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT05788887/Prot_SAP_ICF_001.pdf